CLINICAL TRIAL: NCT03197142
Title: Cardiac Arrest Registry of the Lombardia Region (Lombardia CARe)
Acronym: Lombardia CARe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Azienda Regionale Emergenza Urgenza - AREU Lombardia (Other); Azienda Socio-Sanitaria Territoriale di Pavia (Unknown); Azienda Socio Sanitaria Territoriale di Lodi (Other); Azienda Socio-Sanitaria Territoriale di Crema (Unknown); Azienda Socio Sanitaria Territoriale di Mantova (Other); Azienda Socio Sanitaria Territoriale di Cremona (Other); Azienda Socio-Sanitaria Territoriale Sette Laghi (Unknown); Azienda Socio Sanitaria Territoriale della Valle Olona (Other); Azienda Socio-Sanitaria Territoriale Lariana (Unknown); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); ASST FRANCIACORTA (Unknown); Azienda Socio Sanitaria Territoriale del Garda (Other Government); ASST Valcamonica (Unknown)
Responsible Party: Principal Investigator, Simone Savastano, Cardiologist, Principal Investigator of Pavia CARe, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Lombardia CARe
Record Dates: First submitted 2017-06-17; First posted 2017-06-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: cardiac arrest; resuscitation; Out-Of-Hospital Cardiac Arrest; CPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest: All the patients who suffered an out-of-hospital cardiac arrest in the Lombardia Region

SUMMARY:
The registry enroll all the patients who suffered an out-of-hospital cardiac arrest in the Lombardia Region with a follow-up up to ten years after the event.

DETAILED DESCRIPTION:
The registry is an observational study which enroll all the patients who suffered an out-of-hospital cardiac arrest of any etiology in the Lombardia Region The follow-up of the patients is at 1 month after the event, 6 month and every year up to five years after the event.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest of any etiology in the Lombardia Region

Exclusion Criteria:

* In-hospital cardiac arrest

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who suffered an out-of-hospital cardiac arrest of any etiology in the Lombardia Region
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Survival with good neurological outcome for OHCA patients of any etiology | From cardiac arrest date up to 10 years or up to death, whichever come first
  Survival with Cerebral Performance Category of 1 or 2

CONTACTS AND LOCATIONS:
Locations (21):
- Italy (21):
  - Azienda Socio Sanitaria Territoriale di Crema, Crema, Cremona
  - Azienda Socio Sanitaria Territoriale di Mantova, Mantova, Mantova
  - AAT Brescia, Brescia
  - Fondazione Poliambulanza di Brescia, Brescia
  - Spedali Civili di Brescia, Brescia
  - Ospedale di Busto Arsizio, Gallarate, Busto Arsizio
  - Ospedale Mater Domini di Castellanza, Castellanza
  - AAT Como, Como
  - Ospedale Sant'Anna di Como,Ospedale Sant'Antonio Abate di Cantù e Ospedale Erba-Renaldi di Menaggio, Como
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - AAT 118 - Cremona, AREU Lombardia, Cremona
  - Ospedale di Legnano, Legnano
  - Azienda Socio Sanitaria Territoriale di Lodi, Lodi
  - AAT 118 - Lodi, AREU Lombardia, Lodi
  - AAT 118 - Mantova, AREU Lombardia, Mantova
  - AAT 118 - Pavia, AREU Lombardia, Pavia
  - IRCCS Policlinico San Matteo, Pavia
  - AAT Varese, Varese
  - Ospedale di Angera, Cittiglio, Varese Circolo, Luino, Tradate, Varese
  - Ospedale Civile di Vigevano, Azienda Socio-Sanitaria Territoriale di Pavia, Vigevano
  - Ospedale Civile di Voghera, Azienda Socio-Sanitaria Territoriale di Pavia, Voghera

IPD SHARING:
Plan to Share IPD: No